CLINICAL TRIAL: NCT01458886
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Parallel-group Study Assessing Efficacy and Safety of a 12 Week Treatment With BI 54903 Administered at 90.9 Mcg b.i.d. and 181.8 Mcg q.d. (p.m.Dosing) Via Respimat® Inhaler in Patients With Asthma Inadequately Controlled on Short Acting Beta-2 Agonist (SABA) Therapy Alone
Brief Title: Study on BI 54903 (Inhaled Corticosteroid) Administered Once Daily or Twice Daily Via Respimat Inhaler in Patients With Asthma Inadequately Controlled on Short Acting Beta-2 Agonist (SABA) Therapy Alone
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1248.2; 2010-023165-22 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (3):
- BI 54903 LD b.i.d. (Experimental): Patients receive 2 puffs b.i.d. via Respimat inhaler
  Interventions: Drug: BI 54903
- BI 54903 MD q.d. (Experimental): Patients receive 2 puffs q.d. via Respimat inhaler (p.m.) combined with 2 puffs placebo (a.m.)
  Interventions: Drug: BI 54903 MD; Drug: Placebo matching Respimat
- Placebo (Placebo Comparator): Patients receive 2 puffs b.i.d. via Respimat inhaler
  Interventions: Drug: Placebo matching Respimat

INTERVENTIONS:
Drug: BI 54903 MD — 2 puffs b.i.d. via Respimat inhaler
  Arms: BI 54903 MD q.d.
Drug: Placebo matching Respimat — 2 puffs a.m. via Respimat inhaler
  Arms: BI 54903 MD q.d.
Drug: Placebo matching Respimat — 2 puffs a.m. via Respimat inhaler
  Arms: Placebo
Drug: BI 54903 — 2 puffs LD b.i.d. via Respimat inhaler
  Arms: BI 54903 LD b.i.d.

SUMMARY:
The aim of this study is to assess and compare efficacy and safety of BI 54903 at doses of very low dose twice daily (b.i.d) and low dose once daily (evening dosing) and placebo over an 12-week treatment period in asthmatic patients aged 12 to 65 years inadequately controlled on short acting beta-2 agonist (SABA) therapy alone as demonstrated by a decrease in forced expiratory volume in 1 second (FEV1) (not less than 10 %, and equal to or less than 25%) and an Asthma Control Questionnaire (ACQ-6) of not less than 1.5 at time of randomisation.

ELIGIBILITY:
Inclusion criteria:

To enter run-in following completion of pre-screening period:

1. All patients must sign and date an Informed Consent Form (ICF) at Visit 0 consistent with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) guidelines and local legislation prior to participation in trial, which includes medication washout and restrictions
2. Male and female patients aged at least 12 to 65 years.
3. All patients must have a history of asthma diagnosed by a physician for at least three months at the time of enrolment into the trial according to the 2009 Global Initiative for Asthma (GINA) Guidelines. The initial diagnosis of asthma must have been made before the age of 40 years.
4. All patients must be on a maintenance treatment with either medium-dose inhaled corticosteroids (ICS) plus long acting beta-2 agonist (LABA) or high-dose ICS without LABA, stable for at least six weeks prior to Visit 1.
5. All patients must have a pre-bronchodilator forced expiratory volume in 1 second (FEV1) of not less than 60 to 90% of predicted normal and an Asthma Control Questionnaire (ACQ-6) mean score of less than 1.5 at the pre-screening Visit 1.
6. Patients must be never-smokers or ex-smokers with a smoking history of less than10 pack-years and smoking cessation at least one year prior to screening .
7. Patients must be able to use Respimat® inhaler and metered dosed inhaler (MDI) correctly
8. Patients must be able to perform all trial-related procedures including technically acceptable pulmonary function tests and electronic pear expiratory flow (PEF) measurements, and must be able to maintain records during the study period as required in the protocol.

   To enter treatment period following additional criteria have to be met (at randomisation visit):
9. All patients must have an improvement in FEV1 not less than 12 % above baseline and an absolute change of at least 200 mL within 15-30 min after administration of 400 mcg salbutamol/albuterol hydroflouroalkane (HFA) MDI., as demonstrated at Visit 1 or during one of the visits during the run-in period.
10. During the run-in period (at the same clinic visit) all patients must be both symptomatic (ACQ-6 mean score equal to or greater than 1.5) and have shown a decrease in morning pre-bronchodilator FEV1 not less than 10% and less than or equal to 25% from pre-screening baseline FEV1 at Visit 2.

Exclusion criteria:

1. Patients with significant pulmonary disease other than asthma or other significant medical conditions (as determined by medical history, examination and clinical investigations at screening) that may, in the opinion of the investigator, result in any of the following: (i) put the patient at risk because of participation in this trial or (ii) influence the results of the trial or (iii) cause concern regarding the patient's ability to participate in the trial.
2. Patients with a clinically relevant, abnormal screening haematology and/or blood chemistry finding, if the abnormality indicates a significant disease as defined in exclusion criterion no. 1.
3. Patients with a history of upper or lower respiratory tract infection (URTI/LRTI) in the past four weeks prior to the pre-screening Visit 1, and during pre-screening and run-in periods.
4. Patients with any exacerbation of their underlying asthma during the eight weeks prior to the pre-screening Visit 1.
5. Patients with active allergic rhinitis requiring treatment with systemic corticosteroids.
6. Any of the following criteria are met during the pre-screening / run-in period (Visits 1 - 6):

   1. in clinic pre-bronchodilator FEV1 % predicted less than 40%,
   2. more than 12 puffs rescue salbutamol/albuterol HFA MDI per day for > 2 consecutive days,
   3. exacerbation of asthma.
7. Patients with a history of pneumonectomy or who are planning to undergo thoracotomy for any reason.
8. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the six weeks prior to the first screening visit 1.
9. Patients with two or more hospitalizations for asthma within the previous 12 months.
10. Patients with a recent history of myocardial infarction during the last twelve months or known coronary heart disease that requires treatment
11. Patients with a history of hospitalisation due to heart failure in the past twelve months
12. Patients with myocarditis or any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year
13. Patients with significant alcohol or drug abuse in the opinion of the investigator within the past two years
14. Patients with rheumatoid arthritis or other systemic diseases that require immune system modulating treatment
15. Patients suffering from or with a history of glaucoma, increased intraocular pressure, and/or cataracts
16. Pregnant or nursing women
17. Women of childbearing potential not using a highly effective method of birth control.
18. Patients who have been treated with anti-IgE-antibodies (e.g. omalizumab - Xolair®) or other immune system modulating antibodies such as TNF alpha blockers within six months prior to Visit 1.
19. Patients who have been treated with the following drugs during the past four weeks prior to Visit 1 or are foreseen to need this during the study:

    1. Non-selective ß-blockers (topical cardio-selective beta-blocker eye medications for non-narrow angle glaucoma are allowed),
    2. Oral or other systemic corticosteroids,
    3. Oral beta-agonists,
    4. Changes in allergen desensitisation therapy in last 6 months,
    5. Immune system modulating agents such as methotrexate or cyclosporine,
    6. Inhibitors of cytochrome P450 3A4 such as antifungals (e.g. ketoconazole, itraconazole), antibiotics (e.g. erythromycin) or antiretroviral drugs.
20. Patients who have been treated with leukotriene modifiers, cromones or theophylline within two weeks prior to Visit 1.
21. Patients who have been treated with tiotropium within 3 weeks prior to Visit 1.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Mean change from randomisation baseline to the end of the 12-week treatment period in evening trough (pre-dose and pre-rescue bronchodilator) FEV1 | 12 weeks

SECONDARY OUTCOMES:
Mean change from randomisation baseline to the end of the 12-week treatment period in morning and evening trough (pre-dose and pre-rescue bronchodilator) FVC | 12 weeks
Mean change from randomisation baseline in morning and evening trough (pre-dose and pre-rescue bronchodilator) FEV1 and FVC after 2, 4 and 8-week treatment periods, and in morning trough FEV1 after 12 week treatment period | 12 weeks
Mean pre-dose (and pre-rescue) PEF as assessed via AM2+ device (in the morning and evening) of the last week of the 12-week treatment period | 12 weeks
Mean rescue medication use (daytime and night-time) as assessed via AM2+ device (in the morning and evening) of the last week of the 12-week treatment period | 12 weeks
Asthma control questionnaire (ACQ-6) | 12 weeks
Asthma quality of life questionnaire (AQLQ(S)+12) | 12 weeks
Time to withdrawal due to first asthma exacerbation | 12weeks
Daytime 12-h FEV1 profiles after 12-week treatment period (FEV1 AUC0-12h) | 12 weeks
Mean change from randomisation baseline in morning and evening trough (pre-dose and pre-rescue bronchodilator) FEF25-75 after 2, 4, 8 and 12 week treatment periods | 2, 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim